CLINICAL TRIAL: NCT05730946
Title: Understanding The Challenges and Concerns Faced by Parents of Children With Cleft Lip and/or Palate: A Qualitative Study
Brief Title: Challenges and Concerns Faced by Parents of Children With Cleft Lip and/or Palate
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Alaa Mohammed Yehia, Assistant Lecturer at Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Ain Shams University
Other Study IDs: 1137
Record Dates: First submitted 2023-02-02; First posted 2023-02-16 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Cleft Lip and Palate
Keywords: Cleft Lip and Palate; Challenges; Concerns
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Egyptian parents of cleft lip and/ or palate (CLP) patients: Egyptian parents of CLP patients presented to the cleft lip & palate clinic at Ain Shams university.
  Interventions: Diagnostic Test: Interview- based questionnaire

INTERVENTIONS:
Diagnostic Test: Interview- based questionnaire — Interview-based questionnaire by the use of an interview guide to explore and understand the Challenges faced in the past and the concerns for the future experienced by parents of CLP patients.

SUMMARY:
Cleft lip and/or palate (CLP) are the most common oro-facial congenital anomalies. These anomalies have an impact on feeding, speech and speech development, facial aesthetics & oral health, all of which are factors that heavily impact the quality of life of CLP patients. CLP also has an effect on the families' social and psychological health.

Qualitative research helps understand the perspectives of the participants by exploring the psycho-social aspects of care. Phenomenological approach is a qualitative research method that aims to borrow participants' lived experiences to better understand a specific phenomenon. Currently, there is no clear understanding of the fears, anxieties, and challenges faced by parents of CLP patients in Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Parents of Patients with non-syndromic CLP.

Exclusion Criteria:

* Parents of Patients presenting with dental pain.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Egyptian parents of CLP patients presented to cleft lip & palate clinic at Ain Shams university.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Challenges & concerns faced by the parents of CLP patients | 1 year
  The tool of measurement in the present qualitative study is In-depth interviews utilizing an interview guide (questionnaire).
  The recorded interviews will be transcribed by one of the authors after which thematic data analysis will be conducted. Codes will be developed by two researchers individually and intercoder meetings will held to encourage intercoder reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Mohamed Ali, Prof of PD, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johansson B, Ringsberg KC. Parents' experiences of having a child with cleft lip and palate. J Adv Nurs. 2004 Jul;47(2):165-73. doi: 10.1111/j.1365-2648.2004.03075.x. PMID 15196190
- [Background] Ghirotto L, De Panfilis L, Di Leo S. Health professionals learning qualitative research in their workplace: a focused ethnography. BMC Med Educ. 2020 Aug 17;20(1):269. doi: 10.1186/s12909-020-02191-5. PMID 32807161
- [Background] Baker C, Wuest J, Stern PN. Method slurring: the grounded theory/phenomenology example. J Adv Nurs. 1992 Nov;17(11):1355-60. doi: 10.1111/j.1365-2648.1992.tb01859.x. PMID 1430643
- [Background] Hennink M, Kaiser BN. Sample sizes for saturation in qualitative research: A systematic review of empirical tests. Soc Sci Med. 2022 Jan;292:114523. doi: 10.1016/j.socscimed.2021.114523. Epub 2021 Nov 2. PMID 34785096
- [Background] Turner DW. Qualitative interview design: A practical guide for novice investigators. Qual Rep. 2010;15(3):754-60.
- [Background] Elmouden L, Elgasmi F, Ousehal L. Quality of Life in Adolescents with Cleft Lip and Palate. In: Gülşen A, editor. Current Treatment of Cleft Lip and Palate. 2020.